CLINICAL TRIAL: NCT06885177
Title: TECTONIC CAD Intravascular Lithotripsy (IVL) IDE Study
Brief Title: TECTONIC CAD IVL IDE Study
Acronym: TECTONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10540
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Calcification; Coronary Artery Disease; Stenotic Coronary Lesion
Keywords: Lithotripsy; Coronary Artery Calcification; PCI (Percutaneous Coronary Intervention); De Novo Coronary Arteries
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The study device consists of the IVL Console, a single-use disposable Catheter, and the Integrated Connection Cable with Handpiece.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Abbott Coronary IVL System) (Experimental): Participants will receive treatment with Abbott's Coronary IVL System followed by stenting.
  Interventions: Device: Experimental

INTERVENTIONS:
Device: Experimental — Participants will receive treatment with Abbott's Coronary IVL System followed by stenting.

SUMMARY:
A prospective, single-arm, open-label, multi-center IDE study with up to 55 US sites

DETAILED DESCRIPTION:
The TECTONIC CAD IVL IDE Study is a prospective, single-arm, open-label, multi-center study to evaluate the safety and effectiveness of the Abbott Coronary IVL System to treat severely calcified, stenotic de novo coronary arteries prior to stenting in 335 subjects at up to 55 sites in the US. The clinical outcomes from the study will be compared to pre-specified performance goals (PG) established using medical/scientific literature. This clinical investigation will be conducted under an investigational device exemption (IDE) and is intended to support market approval of the Abbott Coronary IVL System in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must sign and date a written informed consent form before any study-specific tests or procedures are performed.
3. Subject is able and willing to comply with all protocol requirements.
4. Subject has native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI.
5. For subject with unstable ischemic heart disease, cardiac biomarker (troponin) must be less than or equal to the upper reference limit (URL) within 12 hours prior to the procedure.
6. For subject with stable ischemic heart disease, cardiac biomarker (troponin) must be less than or equal to 1.5 times the URL. Blood for cardiac biomarkers may be drawn prior to the procedure or at the time of the procedure from the side port of the sheath.

6a. If drawn prior to the procedure, cardiac biomarker (troponin) must be less than or equal to 1.5x the URL within 12 hours prior to the index procedure.

6b. If drawn at the time of the procedure from the side port of the sheath prior to any intervention, cardiac biomarker results need to be analyzed and resulted prior to registering the subject into the study.

7) Left ventricular ejection fraction (LVEF) ≥ 25% within 6 months (note: in the case of multiple assessments of LVEF, the measurement closest to enrollment will be used for these criteria; may be assessed at time of index procedure).

8) Lesions in non-target vessels requiring PCI may be treated either: a. >30 days prior to the study procedure if the procedure was unsuccessful or complicated; or b. >24 hours prior to the study procedure if the procedure was successful and uncomplicated; or c. >30 days after the study procedure (in 1 or 2 non-target vessels).

Anatomic Inclusion Criteria

Anatomic inclusion criteria are applied at the time of cardiac catheterization for PCI by the investigator and are visually assessed by angiography. The anatomic inclusion criteria include the following:

1. The target lesion must be a single de novo coronary lesion that has not been previously treated with ANY interventional procedure.
2. Single de novo target lesion stenosis of protected left main coronary artery (LMCA), or left anterior descending artery (LAD), right coronary artery (RCA), left circumflex artery (LCX), or ramus intermedius (RI), or of their branches with: a. Stenosis of ≥70% and <100% or b. Stenosis ≥50% and <70% with evidence of ischemia via positive stress test, or fractional flow reserve (FFR) value ≤0.80, or RFR/iFR <0.89 (or any other non-hyperemic pressure index), or IVUS or OCT minimum lumen area ≤4.0 mm^2
3. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm.
4. The lesion length must not exceed 36 mm. 4a) Tandem lesions are allowed and considered one lesion if they are <5 mm apart and as long as the total lesion length does not exceed 36 mm, except for distal lesions without planned treatment and that are in vessels ≤2.0 mm in diameter.
5. The target vessel must have TIMI grade 3 flow at baseline; may be assessed after pre-dilatation.
6. Evidence of calcification at the lesion site by, a. Angiography, with fluoroscopic radiopacities noted as severe (radiopacities noted without cardiac motion before contrast injection compromising both sides of the arterial lumen) OR b. IVUS or OCT, with presence of ≥270 degrees of calcium on at least 1 cross section.
7. Ability to pass a 0.014" guide wire across the lesion.

Exclusion Criteria:

1. Subject has other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results.
2. Subject is a member of a vulnerable population including individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent.
3. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the Primary endpoint. For the purposes of this criterion, "participation" is defined as being registered in another trial.
4. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period. For subjects with childbearing potential, a urine or blood pregnancy test is required within 7 days prior to index procedure to verify that subject is not pregnant. Note: Investigators should instruct female patients of childbearing potential to use safe contraception for 12 months after the procedure (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches, hormonal vaginal devices, injections with prolonged release). It is acceptable to include subjects having a sterilized regular partner.
5. Subject unable to tolerate dual antiplatelet therapy (i.e., aspirin, and either clopidogrel, prasugrel, or ticagrelor) for at least 6 months.
6. Subject has an allergy to imaging contrast media which cannot be adequately pre-medicated.
7. Subject experienced an acute MI (either ST-segment elevation myocardial infarction, STEMI or non-ST-segment elevation myocardial infarction, NSTEMI) within 7 days prior to index procedure, defined as a clinical syndrome consistent with an acute coronary syndrome with troponin or CK- MB greater than 1 times the local laboratory's ULN.
8. Subject has New York Heart Association (NYHA) class III or IV heart failure.
9. Subject has renal failure with serum creatinine >2.5 mg/dL, or chronic dialysis.
10. Subject has a history of a stroke or transient ischemic attack (TIA) within 6 months, or any prior intracranial hemorrhage or permanent neurologic deficit.
11. Subject has an active peptic ulcer or upper gastrointestinal bleeding within 6 months.
12. Subject has an untreated pre-procedural hemoglobin <8 g/dL or intention to refuse blood transfusions if one should become necessary.
13. Subject has a coagulopathy, including but not limited to platelet count <100,000 or International Normalized ratio (INR) >1.7 (INR is only required in subjects who have taken warfarin within 2 weeks of enrollment).
14. Subject has a hypercoagulable disorder such as polycythemia vera, platelet count >750,000 or other disorders.
15. Subject has uncontrolled diabetes defined as a HbA1c ≥10%.
16. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics.
17. Subject in cardiogenic shock or with clinical evidence of left-sided heart failure (S3 gallop, pulmonary rales, oliguria, or hypoxemia).
18. Subject has uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg).
19. Subject with a life expectancy of less than 1 year.
20. Subject has had interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days prior to the index procedure.
21. Subject has planned interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days after the index procedure.
22. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery.
23. Subject has a previous stent in the target vessel implanted within the last year.
24. Planned use of atherectomy, scoring or cutting balloon, ultra-high pressure non-compliant balloon, excimer laser coronary atherectomy (ELCA), drug-coated balloon (DCB) or any investigational device other than the current study device

Anatomic Exclusion Criteria

Anatomic exclusion criteria are applied at the time of cardiac catheterization for PCI by the investigator and are visually assessed by angiography. The anatomic exclusion criteria include the following:

1. Unprotected LMCA diameter stenosis >30%.
2. Target lesion has a myocardial bridge.
3. Target vessel is excessively tortuous, defined as the presence of 2 or more bends >90 degrees or 3 or more bends >75 degrees.
4. Definite or possible thrombus in the target vessel.
5. Evidence of aneurysm in target vessel within 10 mm of the target lesion.
6. Target lesion in ostial location (within 5 mm of the vessel origin) of the LAD, LCX, or RI and per the physician's discretion would require stenting into the LMCA.
7. Target lesion is a bifurcation with the side branch having ostial diameter stenosis ≥50% and is an intervenable target (e.g. ≥2.0mm in diameter).
8. Second lesion with >50% stenosis in the same target vessel as the target lesion, including planned treatment of side branches and distal lesions that are ≥2.0 mm in diameter.
9. Target lesion is located in a native vessel that can only be reached by going through an existing coronary artery bypass graft.
10. Any previous stent within 10 mm of the target lesion.
11. Imaging evidence of a dissection (NHLBI dissection grades D-F) in the target vessel after guide wire passage and/or prior to start of IVL treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Procedural success with final mean residual stenosis <50% and without in-hospital TLF. | Within 48 hour post index procedure or prior to discharge, whichever is earlier.
  The primary effectiveness endpoint is procedural success that is defined as stent delivery with final mean residual stenosis <50% (core laboratory assessed) and without in-hospital TLF.
Primary Safety Endpoint: TLF at 30-days post index procedure | 30-days post index procedure
  The primary safety endpoint is TLF (Target lesion failure) defined as a composite of Cardiac Death, TV-MI (Target vessel myocardial infarction), which includes peri-procedural myocardial infarction (PPMI) defined by ARC-2 and spontaneous MI defined by the fourth universal definition of MI (UDMI), and CD-TLR (clinically driven target lesion revascularization)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - HonorHealth, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Kaiser Permanente - San Francisco, San Francisco, California
  - ClinRé 001-100 - Denver, Denver, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The Cardiac & Vascular Institute Research Foundation, LLC, Gainesville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Mayo Clinic of Jacksonville, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Mt. Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Wellstar Kennestone Regional Medical Center, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Bryan Heart, Lincoln, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ascension St. John Jane Phillips, Bartlesville, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health System, Mechanicsburg, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Baylor Scott & White Heart & Vascular Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Shannon Clinic, San Angelo, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No